CLINICAL TRIAL: NCT04335825
Title: Surgical and Refractive Outcomes of Combined Phaco-ExPress Versus Phacotrabeculectomy - 6 Months Results.
Brief Title: Surgical and Refractive Outcomes of Combined Glaucoma Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1774
Record Dates: First submitted 2020-03-28; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma; Ocular Hypertension; Filtering Surgery
Keywords: glaucoma combined surgery; postoperative astigmatism; postsurgery refractive error
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phacotrabeculectomy (Active Comparator): patients undergoing phacotrabeculectomy
  Interventions: Procedure: phacotrabeculectomy
- ExPress device implantation (Active Comparator): patients undergoing ExPress antiglaucoma surgery combined with phacoemulsification
  Interventions: Procedure: ExPress antiglaucoma surgery combined with phacoemulsification

INTERVENTIONS:
Procedure: phacotrabeculectomy — combined antiglaucoma procedure: trabeculectomy with phacoemulsification
  Arms: phacotrabeculectomy
Procedure: ExPress antiglaucoma surgery combined with phacoemulsification — combined antiglaucoma procedure: ExPress device implantation with phacoemulsification
  Arms: ExPress device implantation

SUMMARY:
The aim of the study is to examine surgical and refractive outcomes of glaucoma combined surgery in six months period of follow up

DETAILED DESCRIPTION:
Trabeculectomy and implantation of the Ex-Press device belong to the same group of anti-glaucoma procedures improving subconjunctival outflow. The most frequently performed glaucoma surgery of choice is still trabeculectomy, although the less invasive implantation of the Ex-Press device is also an effective alternative. Despite the wide application of these two techniques, their impact on postoperative refraction is not entirely known. Quite often, in the early postoperative period there is a decrease in visual function, which is short-term, although there are reports that it can last up to a year after surgery. It can be caused by a reduction in IOP, as well as the direct effect of trabeculectomy on corneal topography, and thus on postoperative astigmatism and refractive error. The occurrence of astigmatism after trabeculectomy has been widely documented Combined operations of implanting the ExPress implant with cataract phacoemulsification differ from phacotrabeculectomy in that, they do not require cutting of the sclera, cutting the limbus and using a punch.

The purpose of our research was to compare the phacotrabeculectomy and phacoemulsification combined with Express device implantation in terms of incidence of postoperative astigmatism in a prospective randomized study, and to attempt to determine what factors determine its size.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma with coexisting cataract graded Nuclear-Cortical 1 (NC1) and Nuclear-Cortical 2 (NC2), according to the The Lens Opacities Classification System III (LOCS III scale), was an indication for surgery.
* Patients with primary open-angle glaucoma (POAG), pseudoexfoliation glaucoma (PXG) and pigmentary glaucoma (PG), in which satisfactory intraocular pressure (IOP >21 mmHg) was not achieved despite maximally-tolerated topical and systemic medication, were qualified for treatment.
* Additional inclusion criteria were as follows: well documented progression of visual field defects, significant diurnal variations in the IOP, poor patient compliance, and allergy to topical drugs.

Exclusion Criteria:

* Lack of consent to participate in the study,
* History of eye surgery or laser procedures within the eye,
* Closed or narrow angle glaucoma,
* Diabetes,
* Advanced macular degeneration
* Active inflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
IOP | baseline and six months after surgery
  the change in the level of intraocular pressure

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | baseline and six months after surgery
  the change in the best corrected visual acuity
astigmatism | baseline and six months after surgery
  the change in the value of astigmatism with the use of autokeratorefractometer before and after surgery

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of each participant will be available upon email request for all primary and secondary outcome measures
Supporting Information: Study Protocol
Time Frame: Data will be available on email request for six months after completing the study
Access Criteria: e mail request, after Data Access Agreement is sign

REFERENCES:
- [Result] Chan HHL, Kong YXG. Glaucoma surgery and induced astigmatism: a systematic review. Eye Vis (Lond). 2017 Nov 17;4:27. doi: 10.1186/s40662-017-0090-x. eCollection 2017. PMID 29177182
- [Result] Hong YJ, Choe CM, Lee YG, Chung HS, Kim HK. The effect of mitomycin-C on postoperative corneal astigmatism in trabeculectomy and a triple procedure. Ophthalmic Surg Lasers. 1998 Jun;29(6):484-9. PMID 9640570
- [Result] Alvani A, Pakravan M, Esfandiari H, Safi S, Yaseri M, Pakravan P. Ocular Biometric Changes after Trabeculectomy. J Ophthalmic Vis Res. 2016 Jul-Sep;11(3):296-303. doi: 10.4103/2008-322X.188399. PMID 27621788